CLINICAL TRIAL: NCT02424695
Title: Effects of Gabapentin Enacarbil on Intensity of Cortical Arousal, Heart Rate, Blood Pressure and Anterior Tibialis EMG Responses Associated With PLMs During Sleep in Patients With RLS Using a Novel Computer Assisted Scoring System
Brief Title: Effects of Gabapentin Enacarbil on Arousals, Heart Rate, Blood Pressure and PLMs in Restless Legs Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cleveland Sleep Research Center (Other)
Collaborators: XenoPort, Inc. (Industry); YRT Limited (Unknown)
Responsible Party: Principal Investigator, Mansoor Ahmed M.D., Medical Director, Cleveland Sleep Research Center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: XP-IIT-0031
Record Dates: First submitted 2015-04-15; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Restless Legs Syndrome
Keywords: Cortical arousal intensity; RLS; Heart rate; Blood pressure; PLMs
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid; Gabapentin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Gabapentin Enacarbil Arm (Experimental): Gabapentin Enacarbil (Gen) 600 mg will be administered once daily for 4 weeks
  Matching placebo will be administered once daily for one week prior initiation of treatment with GEn
  Interventions: Drug: Gabapentin Enacarbil (GEn); Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin Enacarbil (GEn) — HORIZANT Extended-Release Tablets containing 600 mg of gabapentin enacarbil are white to off-white, with occasional black/grey spots, oval-shaped tablets debossed with "GS LFG", supplied as:
  600 mg: NDC 53451-0101-1.The drug will be stored at 25°C (77°F) (excursions permitted 15° to 30°C (59° to 86°F)) Matching placebo will be provided by Xenoport Inc.
  Other Names: HORIZANT
Drug: Placebo

SUMMARY:
This is a phase IV single-blind, placebo run-in fixed dose single-group study to assess objective and subjective effects of GEn on sleep EEG, BP, and anterior tibialis EMG responsivity in patients with RLS. The study will include 8 visits over a period of up to 8 weeks for eligible subjects including a 1 to 3-week Screening/Washout Period, a 1-week placebo run-in period, and a 4-week Treatment Period.The first placebo dose will be administered within 1 to 3 weeks after Screening/Washout. The total duration of the study from the first subject enrolled to the last subject completed will be approximately 1 year.

DETAILED DESCRIPTION:
Evidence from the Sleep Heart Health Study suggests that nocturnal arousals from sleep impact heart rate variability and sleep disorders associated with frequent nocturnal arousals, including restless legs syndrome (RLS), increase the risks of developing cardiovascular disease. The majority of RLS patients, once asleep, exhibit frequent periodic limb movements (PLMs), which cause electroencephalographic (EEG) arousals and sleep fragmentation resulting in poor quality of sleep and daytime consequences. PLMs are also reported to increase heart rate.The precise nature of the relationship between PLMs and their impact on heart rate and blood pressure is not clear. This may relate to the fact that PLMs are scored as either present or absent and without accounting for the differences in intensity of muscle activity during individual PLMs and intensity of associated arousals. In fact PLMs have been reported to vary from barely visible to very intense changes in the anterior tibialis electromyogram (EMG). This study will evaluate the effects of gabapentin encarbil (GEn) on intensity of cortical arousals associated with PLMs using a newly developed computer assisted scoring system which allows for scaling microarousals in the EEG. The anterior tibialis EMG intensity, continuous blood pressure and heart rate will be measured.

The study design is a phase IV single center, single blind, placebo run-in fixed dose single group study in twenty subjects with moderate to severe restless leg syndrome. It includes a one- three week screening washout period, one week of placebo run-in and four- week treatment period with GEn 600 mg once daily. Subjects will be instructed to take their study medication once daily with food in the evening at approximately 5 PM. If the dose is not taken at the recommended time, the next dose should be taken the following day at the regularly scheduled time (about 5 PM the next evening). Subjects will be blinded to treatment (placebo versus active drug).

Polysomnography (PSG) will be obtained for two nights of baseline at the end of placebo run-in and at the end of four weeks of treatment with gabapentin encarbil 600 mg. Medical history and cardiovascular risk factors will be assessed at Screening. RLS disease history, previous/current RLS therapy, augmentation history and evidence of sleep disturbance will be obtained.Severity of RLS will be determined using the International Restless Legs Syndrome (IRLS) scale. The Berlin questionnaire will be used to identify the risk (low to high) of sleep disordered breathing. The Beck Depression Inventory (BDI-II) will be administered to identify depression and its severity at Screening. Electrocardiogram (ECG), clinical laboratory test and urine pregnancy test will be conducted at Screening to determine eligibility. Also to determine eligibility, subjective evidence of sleep disturbance will be assessed per daily sleep diary at Visit 2. A physical exam will be performed at the beginning of the Placebo Run-in Period.

The visit schedule includes: Screening; Scheduled Tests/Exams; Placebo administration visit; Baseline PSG visits; Baseline Visit; End of treatment PSG visits; Adverse Event Evaluation (for all subjects);Unscheduled clinical evaluation visit; and End of Study Visit.

Primary outcome will involve change from baseline (end of run-in period) in cortical arousal intensity associated with PLMs for subjects treated with Gen 600 mg QD for 4 weeks. PSG studies will be recorded for 8 hours using standard techniques described by R&K. Cortical EEG arousals will be scored using wavelet analysis of C3/A2 and C4/A1 EEG signals. Arousals scored in NREM sleep will be assigned a score from 0-9. This arousal scaling is entirely subjective. Wavelet analysis will be performed on each of the scaled arousals using wavelet features that correlate with arousal intensity. The arousal intensity will be measured using Wavelet Transform which is superior for analyzing signals such as EEG.

Beat to beat heart rate measurement will identify the highest value in the interval 2-12 seconds preceding each arousal which will be used as a baseline heart rate. The highest heart rate in the interval between arousal and at 8 seconds after its end, and the difference from baseline will represent the change in heart rate associated with the arousal.

Blood pressure changes will be identified using the same technique as the heart rate changes. Continuous blood pressure will be monitored using Somnotouch RESP. Using the 2-12 seconds preceding each arousal, any identified change between onset of arousal and at 8 seconds after its end will represent the change in blood pressure.

PLM intensity will be derived by measuring the highest anterior tibialis EMG amplitude during the 2-12 seconds prior to arousal onset and comparing to maximum EMG amplitude during PLMs with or without associated arousal.

The Rechtschaffen and Kales (R&K) standard PSG parameters include: TST (total sleep time), WASO (wake after sleep onset), LPS10 (latency to persistent sleep), SE (sleep efficiency), Awakenings Index (number of awakenings per hour of sleep), AI (arousals index), sleep stage percentages, PLMI (periodic limb movements per hour), and PLMAI (periodic limb movements associated with arousal per hour).

The secondary subjective efficacy endpoints are: 1) the mean change from Baseline to the end of the Treatment Period in International Restless Legs Syndrome (IRLS) Rating Scale total score, (2) proportion of responders ("much"/ "very much" improved) on the investigator-rated Clinical Global Impression-Improvement (CGI-I) scale, and proportion of responders ("moderately better" to "a great deal better") on the Patient Global Impression of Change (PGIC) scale (4) the mean change from baseline to the end of the Treatment Period in PSQ, SSQ items, RLSQoL, RLS-NDI and ESS scores

The IRLSSG has developed and validated a 10-item scale for assessing the severity of RLS. The IRLS Rating scale will be assessed at the screening visit, the placebo initiation visit, the baseline visit and end of study visit (and at the ET visit for subjects who withdraw prematurely). The investigator-rated CGI-I will be recorded at Baseline (end of placebo administration) and at the end of the Treatment Period and at the ET visit, if applicable.

The PSQ is a self-rated questionnaire which assesses sleep quality and sleep disturbances over a one month time interval. The RLSQoL is an 18-item scale that assesses the impact of RLS on daily life, emotional wellbeing, social life, and work life. The ESS is an assessment used to measure average longtime sleepiness whereby subjects self-rate questions on how likely they are to fall asleep in eight different situations. The PSQ, RLSQoL and ESS will be recorded at Baseline and at the end of the Treatment Period and at the ET visit, if applicable.

The SSQ is a daily sleep diary where subjects record their sleep activities and report the quality of their sleep over the past 24 hours on an 11 point numeric rating scale ranging from 0 ("very poor") to 10 ("excellent"). The RLS-NDI measures the impacts of RLS on next day functioning. The impacts include activities of daily living (i.e., work, household chores), cognitive functioning (i.e., concentration, forgetfulness, mental tiredness, alertness), emotional functioning (i.e., irritability, depressed mood), physical functioning (i.e., physical tiredness, active leisure activities), energy, daytime sleepiness, and social functioning (i.e., relationships, social activities/situations). The final measure consists of 14 items assessed "today" and rated on a numeric rating scale. Subjects will be instructed to complete the daily diary and the RLS-NDI over the 7 days preceding Visit 4 (PSG 2 visit) and Visit 7 (PSG 4 visit).

The following safety assessments will be performed during this study:

Physical examination, including height as with other screening only measurements; Weight measurements;Vital sign measurements, including blood pressure and pulse rate;Pregnancy testing; AE reporting;ECG (for screening only); Laboratory safety tests (at screening)

The primary efficacy endpoint is the reduction from placebo-baseline in cortical arousal intensity associated with PLMs after treatment with GEn. A sample size of 20 subjects is estimated by a priori power analysis (G*Power 3.1.9.2) to achieve 92% power for a 2-sided 5% paired t-test with an effect size of 0.80. The primary efficacy analysis will be performed on the per-protocol population who completed the study taking 600 mg GEn/day of the study drug. For subjects who prematurely withdraw from the study, EOS PSG will be acquired provided they received at least 2 weeks of treatment with GEn. All data for primary and secondary endpoints will be analyzed using a paired t-test. 95% confidence intervals will be provided for the true mean treatment difference. Descriptive statistics will be reported for the primary and secondary endpoints by placebo-baseline visit and treatment group. To further evaluate treatment effects, the association between the changes from baseline in primary objective and secondary subjective endpoints will be evaluated using Pearson correlation coefficients. Safety and tolerability analyses will focus primarily on frequency of treatment emergent adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ages 18 to 65 years with a diagnosis of primary moderate to severe RLS
2. A minimum of 6-month history of RLS symptoms
3. IRLS score >15 points (at visits 1 and 2) and a score of > 2 on item 4
4. RLS symptoms on at least 15 days during the month prior to screening (or if on treatment, similar symptom frequency before the start of treatment)
5. RLS symptoms for >4 out of 7 evenings /day during the week prior to screening
6. History of sleep disturbance due to RLS over the last 3 months
7. Subjective history of WASO ≥ 60 min; TST < 6.5 hours; subjective sleep latency ≥ 30 min on at least 3 nights per week within the last 3 months
8. Subjective complaint of WASO ≥ 60 min; TST< 6.5 hours; subjective sleep latency ≥ 30 min on at least 3 nights out of 7on the SSQ during the 1 week prior to Visit 2
9. Objective WASO of ≥30 minutes, TST < 6.5 hours and PLMI ≥ 10 during adaptation in baseline PSG 1
10. Females of child bearing potential willing to use birth control
11. Subject can read understand and sign consent form
12. Subject able to complete the study and to comply with study instructions and procedures

Exclusion Criteria:

1. Subject has an apnea-hypopnea index of ≥10/ hour during adaptation/baseline night PSGs. Subjects with OSA controlled by CPAP will be accepted
2. Evidence of secondary RLS
3. Subject has any of the following medical conditions, laboratory abnormalities or disorders:

   Hepatic impairment Impaired renal function or renal dysfunction requiring hemodialysis; Serum ferritin level <20 mcg/L (ng/mL)
4. Clinically significant ECG abnormalities
5. Any unstable medical condition that could impact subject's safety and study outcomes
6. Uncontrolled hypertension at Screening or at time of treatment initiation
7. Subjects diagnosed with additional sleep disorders other than RLS-associated sleep disturbance
8. Neurologic disease or movement disorder, rheumatoid arthritis, fibromyalgia, uncontrolled psychiatric illness, current diagnosis or history of epilepsy or seizure disorder
9. Chronic hepatitis B or hepatitis C
10. Subject currently suffering from moderate or severe depression
11. Subject unable to discontinue prohibited medications during the Screening period and throughout the duration of the study.
12. Subject has consumed food or beverages containing more than 400 mg of caffeine or other xanthines (e.g., coffee, cola, tea, chocolate) per day over the preceding month prior to Screening or unwilling to refrain from consuming any caffeinated food or beverage within 8 hours prior to any PSG assessment.
13. Subject has typical consumption of >14 alcoholic units in any week, or more than 5 alcoholic units in any single day, over the month preceding the Screening visit or unwilling to refrain from consuming alcohol within 24 hours of any PSG assessment
14. Night workers, shift workers or any others whose sleeping habits are incompatible with the study design, or who would be required to make significant changes to their bedtime during the course of the study
15. Subject who might be non-compliant with the visit schedule, procedures, or medication administration
16. Subject is a pregnant or nursing female
17. A history of allergy or medically significant adverse reaction or intolerance to gabapentin or GEn
18. A history of alcohol, narcotic, benzodiazepine, or other substance abuse or dependence within the past year
19. A history of augmentation or early morning rebound of RLS symptoms without a history of prior response to treatment.
20. Subject has received previous treatment with levodopa/carbidopa, dopamine agonists, pregabalin, gabapentin or GEn in the 3 weeks prior to Visit
21. Subject has received' other treatments for RLS (e.g., opioids, benzodiazepines) at least 2 weeks prior to Visit 2
22. Participation in any clinical drug or device trial within 30 days prior to Baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The mean change from baseline to week 4 in intensity of cortical arousals associated with periodic limb movements (PLMs) | 4 weeks
  Cortical EEG arousals will be scored using wavelet analysis of C3/A2 and C4/A1 EEG signals. Arousals scored in NREM sleep will be assigned a score from 0-9. This arousal scaling is entirely subjective. Wavelet analysis will be performed on each of the scaled arousals using wavelet features that correlate with arousal intensity. The arousal intensity will be measured using Wavelet Transform which is superior for analyzing signals such as EEG.

SECONDARY OUTCOMES:
The mean change from baseline to week 4 in heart rate variability associated with arousals secondary to periodic limb movements (PLMs) | 4 weeks
  Beat to beat heart rate measurement will identify the highest value in the interval 2-12 seconds preceding each arousal which will be used as a baseline heart rate. The highest heart rate in the interval between arousal and at 8 seconds after its end, and the difference from baseline will represent the change in heart rate associated with the arousal.
The mean change from baseline to week 4 in blood pressure associated with arousals secondary to periodic limb movements (PLMs) | 4 weeks
  Blood pressure changes will be identified using the same technique as the heart rate changes. Continuous blood pressure will be monitored using Somnotouch RESP. Using the 2-12 seconds preceding each arousal, any identified change between onset of arousal and at 8 seconds after its end will represent the change in blood pressure.
The mean change from baseline to week 4 in periodic limb movement (PLM) intensity | 4 weeks
  Periodic limb movement (PLM) intensity will be derived by measuring the highest anterior tibialis EMG amplitude during the 2-12 seconds prior to arousal onset and comparing to maximum EMG amplitude during PLMs with or without associated arousal.
The mean change from Baseline to week 4 in Rechtschaffen and Kales polysomnography parameters | 4 weeks
  Polysomnography (PSG) studies will be recorded for 8 hours using standard techniques described by Rechtschaffen and Kales (R&K). The R&K standard PSG parameters include: Total sleep time (TST), wake after sleep onset (WASO), latency to persistent sleep (LPS 10), sleep efficiency (SE), number of awakenings per hour of sleep (Awakenings Index), arousals index (AI), sleep stage percentages, periodic limb movements per hour (PLMI), and periodic limb movements associated with arousal per hour (PLMAI).
The mean change from baseline to week 4 in International Restless Legs Syndrome (IRLS) Rating Scale total score | 4 weeks
The mean change from Baseline to week 4 in proportion of responders ("much"/ "very much" improved) on the investigator-rated Clinical Global Impression-Improvement (CGI-I) scale | 4 weeks
The mean change from Baseline to week 4 in proportion of responders ("moderately better" to "a great deal better") on the patient Global Impression of Change (PGIC) scale | 4 weeks
The mean change from Baseline to week 4 in Post Sleep Questionnaire (PSQ)scores | 4 weeks
The mean change from Baseline to week 4 in Subjective Sleep Questionnaire (SSQ) scores | 4 weeks
The mean change from Baseline to week 4 in Restless Legs Syndrome Quality of Life Questionnaire (RLSQoL) scores | 4 weeks
The mean change from Baseline to week 4 in Restless Legs Syndrome- Next Day Impact Questionnaire (RLS-NDI) scores | 4 weeks
The mean change from Baseline to week 4 in the Epworth Sleepiness Scale (ESS) scores | 4 weeks
Number of subjects with treatment emergent adverse events | 4 weeks
Number of subjects with mild, moderate and severe adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor Ahmed, MD, Principal Investigator — Cleveland Sleep Research Center
Locations (1):
- Cleveland Sleep Research Center, Middleburg Heights, Ohio, United States

REFERENCES:
- [Result] Winkelman JW, Shahar E, Sharief I, Gottlieb DJ. Association of restless legs syndrome and cardiovascular disease in the Sleep Heart Health Study. Neurology. 2008 Jan 1;70(1):35-42. doi: 10.1212/01.wnl.0000287072.93277.c9. PMID 18166705
- [Result] Alessandria M, Provini F. Periodic Limb Movements during Sleep: A New Sleep-Related Cardiovascular Risk Factor? Front Neurol. 2013 Aug 12;4:116. doi: 10.3389/fneur.2013.00116. eCollection 2013. PMID 23964267
- [Result] Walters AS, Rye DB. Review of the relationship of restless legs syndrome and periodic limb movements in sleep to hypertension, heart disease, and stroke. Sleep. 2009 May;32(5):589-97. doi: 10.1093/sleep/32.5.589. PMID 19480225
- [Result] Sforza E, Jouny C, Ibanez V. Time course of arousal response during periodic leg movements in patients with periodic leg movements and restless legs syndrome. Clin Neurophysiol. 2003 Jun;114(6):1116-24. doi: 10.1016/s1388-2457(03)00077-4. PMID 12804680
- [Result] Earley CJ, Silber MH. Restless legs syndrome: understanding its consequences and the need for better treatment. Sleep Med. 2010 Oct;11(9):807-15. doi: 10.1016/j.sleep.2010.07.007. PMID 20817595